CLINICAL TRIAL: NCT06904521
Title: One Health Baseline Research Study
Brief Title: OH Baseline Research Study
Acronym: OHS
Status: Active, not recruiting | Type: Observational
Sponsor: Centre for Infectious Disease Research in Zambia (Other)
Responsible Party: Sponsor
Other Study IDs: 5849-2024; No Identifier was Issued (Other: Sustainable Food Systems Ireland (SFSI) Consortium)
Record Dates: First submitted 2025-03-11; First posted 2025-04-01 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: no Condition, Basic Science
Keywords: One Health

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The One Health baseline research study is essential to comprehensively understand human, animal, and environmental health interrelation within Zambia's diverse ecosystems. The rationale for this study is grounded in three key factors: Firstly, Zambia faces significant health challenges due to zoonotic diseases, which account for a considerable proportion of public health threats. This study aims to gather insights into the knowledge and practices of various system actors regarding food safety, animal disease surveillance, animal medicines controls, and one health systems regulation to provide critical data that will inform targeted interventions and policies. This research aligns with programmed activities under Zambia's National One Health Strategy 2022-2026.

Secondly, the agricultural sector, which is a cornerstone of Zambia's rural economy, heavily relies on healthy livestock and sustainable farming practices. The study will gather insights on the practices of food producers, traders, and markets, essential for the identification of potential areas of improvement and innovation. This is particularly crucial as the agricultural sector supports the livelihoods of a large portion of the population and plays a vital role in food security.

Thirdly, the One Health approach emphasises the importance of collaboration between various sectors and disciplines. This baseline study aims to ascertain levels of awareness among health professionals, veterinarians, environmental scientists, and policymakers. The data collected will serve as a foundation for future research and intervention strategies, ultimately aiming to reduce the incidence of zoonotic diseases and improve overall health outcomes.

DETAILED DESCRIPTION:
1. Introduction Small and medium-scale farmers in Zambia are essential to the agricultural industry, significantly impacting food security and the economy. Typically, small-scale farmers handle less than 5 hectares, concentrating on subsistence farming and local markets. In contrast, medium-scale farmers, who manage between 5 and 20 hectares, participate in subsistence and commercial agriculture.

   The central regulatory bodies overseeing these farmers are the Ministry of Agriculture (MoA), the Ministry of Fisheries and Livestock (MFL), and the Ministry of Green Economy and Environment (MGEE), among others.

   Zambia's provinces provide diverse agricultural opportunities. Agriculture dominates Central, Eastern, and Southern provinces, mainly through smallholder farmers focused on crops, livestock, and horticulture. Luapula, Muchinga, and Northern provinces excel in producing rice, cassava, and vegetables due to favourable agro-ecological conditions. In contrast, North-Western and Western provinces excel in livestock production, playing a crucial role in the nation's meat and dairy sectors. The Copperbelt and Lusaka provinces also feature a mix of commercial and smallholder farming operations, representing Zambia's vibrant agricultural environment. Small and medium-scale farmers throughout these provinces are essential in developing the country's food systems and promoting rural development.

   The food supply chain in Zambia includes smallholder farmers, agricultural businesses, food processors, wholesalers, and retailers. Farmers grow crops and raise livestock, while buyers purchase these products for processing or export. Retailers, from supermarkets to vendors, provide food access for consumers in urban and rural areas. This network is vital for a sustainable food supply chain, supporting livelihoods and ensuring food security in Zambia.
2. Justification of Study The study aimed to gather evidence to support interventions aligned with the global health initiatives and the UN Sustainable Development Goals (SDGs), particularly those related to good health and well-being, zero hunger, and sustainable agriculture. Therefore, conducting this One Health baseline research study was justified by addressing pressing public health concerns, supporting the agricultural sector, promoting interdisciplinary collaboration, and contributing to national and global health objectives. The insights gathered will be instrumental in shaping effective health interventions and policies, ultimately enhancing the well-being of communities across Zambia.
3. Research Question What knowledge do food system actors in Zambia have about One Health principles, including food safety, animal disease surveillance, controls on animal medicine, waste management, and plant health, as well as the regulatory systems for food safety and plant and animal health? The food system actors in the context of this study included a diverse group of stakeholders integral to Zambia's food safety and public health. This included small and medium-scale farmers who are primary producers (farmers producing food of animal and non-animal origin), food producers who may engage in on-farm food processing or operate as standalone processors, traders, and market operators in both formal and informal settings that facilitate the distribution and sale of food products, as well as regional regulators who oversee the enforcement of laws and standards related to food safety, plant health, and animal health.
4. Study Aim and Objectives Aim The research focused on collecting insights regarding knowledge and practices related to food safety, animal disease surveillance, control of animal medicines, and regulation of one health system.

Objectives

* To assess the understanding of small and medium-scale farmers about food safety and plant and animal health, including knowledge of animal medicines.
* To assess the food safety protocols of food manufacturers, which encompass both on-farm and standalone processors.
* To evaluate how traders and markets, both formal and informal, ensure food safety, animal and plant health, and manage waste.
* To assess the knowledge of local inspectors on enforcing legal requirements for waste management, food safety, and plant and animal health, including disease preparedness and animal treatments.

ELIGIBILITY:
Inclusion Criteria:

* Food system actors

Exclusion Criteria:

* Non food system actors

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Food system actors that function along the food supply chain, i.e., Farmers, Food processors, Food buyers, Informal and formal traders and regulators
Sampling Method: Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of food system actors who have knowledge and conduct practices related to food safety, animal disease surveillance, control of animal medicines, and regulation of one health system. | Up to 6 months
  Through the use of quantitative and qualitative interviews, we will gather insights regarding knowledge and practices related to food safety, animal disease surveillance, control of animal medicines, and regulation of one health system.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Riblet, PhD, Principal Investigator — Sustainable Food Systems Ireland; Paula BarryWalsh, Veterinary Doctor, Principal Investigator — Sustainable Food Systems Ireland
Locations (1):
- Centre for Infectious Disease Research in Zambia, Lusaka, Lusaka Province, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified raw participant data will be shared with our funders.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 1st April 2025
Access Criteria: Sustainable Food Systems Ireland (SFSI) Consortium